CLINICAL TRIAL: NCT03766542
Title: Optimal Positive Airway Pressure in Overlap Syndrome: a Randomized Controlled Trial
Brief Title: Continuous Positive Pressure Versus Bi-level in Overlap Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Sao Joao (Other)
Collaborators: Marta Drummond MD PhD (Unknown); Joao Carlos Winck MD PhD (Unknown); Mafalda van Zeller MD Phstud (Unknown)
Responsible Party: Principal Investigator, Miguel R. Goncalves, Clinical Professor, Hospital Sao Joao
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSPAP study
Record Dates: First submitted 2017-02-08; First posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Overlap Syndrome; Nocturnal Hypoventilation
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP (Active Comparator): Oronasal CPAP therapy applied as per current international guidelines
  Interventions: Device: continuous positive airway pressure without ventilatory support
- Bi-level (Experimental): Oronasal Bi-level therapy + supplemental oxygen (if necessary) applied as per current international guidelines
  Interventions: Device: Bi-level positive airway pressure with ventilatory support

INTERVENTIONS:
Device: Bi-level positive airway pressure with ventilatory support — Positive airway pressure will be applied in the experimental group through a oronasal interface, in ventilatory support mode (Bi-level) with a fixed backup rate.
  Arms: Bi-level
Device: continuous positive airway pressure without ventilatory support — Continuous positive airway pressure (CPAP) will be applied in the active comparator group through a oronasal interface.
  Arms: CPAP

SUMMARY:
Continuous positive airway pressure (CPAP) became the established treatment for overlap syndrome (OS). It has been showed that the survival benefits of CPAP favored hypercapnic patients. When considering hypercapnic stable COPD patients, survival benefits occurred when the use of bi- level ventilation therapy was targeted to significantly reduce hypercapnia.

This highlights the relevance of hypercapnia and hypoventilation correction. Thus, the purpose of this study is to compare the use of CPAP to Bi-level ventilation in hypercapnic OS patients, since the later may correct not only the airway patency but also increase the magnitude of each breath.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) and chronic obstructive pulmonary disease (COPD) represent two of the most prevalent respiratory disorders in clinical practice and their coexistence is often described has "overlap syndrome" (OS) In patients with COPD, the coexistence of OSA is associated with an increased risk of death from any cause, and hospitalization because of COPD exacerbation. Treatment with continuous positive airway pressure (CPAP) has been showed to be effective and associated with improved survival and decreased hospitalizations. When CPAP became established treatment for overlap syndrome, a multivariate analysis revealed that the hours of CPAP use were an independent predictor of mortality. Furthermore, it has been showed that the survival benefit of CPAP favors hypercapnic patients with overlap syndrome.

Regarding hypercapnic stable COPD patients, the best results with long-term non-invasive positive pressure ventilation have been noted in studies using more intensive strategies of ventilation, with higher inspiratory pressures and higher backup rates that improved or even normalized daytime hypercapnia. In fact, survival benefits occurred when ventilation was targeted to significantly reduce hypercapnia.

As for typical COPD, overlap syndrome patients might also benefit from optimal daytime hypercapnia correction, which could be better achieved using bi-level ventilation instead of CPAP, since it could not only maintain airway patency but also improve alveolar ventilation.

This study aims to compare CPAP therapy to bi-level ventilatory support in overlap syndrome patients, not only for the efficacy to achieve hypercapnia reduction, but also regarding acute disease exacerbations, symptoms and treatment compliance. Therefore, the authors designed a randomized controlled trial with recruitment and power calculations based on the applicant's own data.

After the diagnosis, patients will be randomized either for CPAP or BPAP treatment.

If CPAP is to be initiated, optimal pressure to maintain upper airway patency will be determined. If there are continued obstructive respiratory events at 15 cm H2O of CPAP, patients will cross-over to the BPAP study arm.

Regarding BPAP titration, patients will be treated with ventilators set in pressure support spontaneous/timed mode, both inspiratory and expiratory positive airway pressures (IPAP and EPAP) will be manually titrated. EPAP will ensure optimal pressure for maintaining upper airway patency and IPAP will be defined according to patient tolerance and pressure support necessary to achieve normal PaCO2 values or to reduce baseline PaCO2 by 20% or more; Follow-up will be performed at 1, 6 and 12 months. Follow-up will include clinical evaluation with physical examination and questionnaires (COPD Assessment test, Epworth Sleepiness Scale and MRC dyspnea score), blood gas analysis, treatment adherence, AHI, nocturnal pulse oximetry and exacerbations.

12-month follow-up will also include lung function test, 6-min walking test and nocturnal capnography.

ELIGIBILITY:
Inclusion Criteria:

* COPD (FEV1/FVC < 70 (post-BD) and history of smoking - 10 PPY)
* FEV1< 80% and COPD symptoms
* AHI ≥ 15 events/hour

Exclusion Criteria:

* Persistent hypercapnic respiratory failure with acidosis (defined as pH <7.30 after bronchodilators)
* Hypoxia requiring long term oxygen therapy
* BMI > 35 kg/m2
* Previously-initiated long term non-invasive positive pressure ventilation
* Other lung disease resulting in respiratory symptoms
* Age <40 years
* Pregnancy
* Malignant comorbidities
* Patients undergoing renal replacement therapy
* Restrictive lung disease causing hypercapnia
* Severe heart failure, unstable angina and severe arrhythmias
* Inability to comply with the protocol

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
diurnal hypercapnia (pCO2 <= 45 mmH2O ) | 1 year
  (PaCO2 <= 45 mmH2O )
nocturnal oxygen desaturation correction | 1 year
  Mean nocturnal SpO2 >=90%, with <10% of the total recording time <90% after correction of leaks)

SECONDARY OUTCOMES:
Changes in FEV1 | 1 year
  Forced Expiratory Volume (FEV1) in first second (% of predicted) from pre-intervention to follow up
Changes in FVC | 1 year
  Forced vital capacity (FVC) (% of predicted) from pre-intervention to follow up
Changes in RV | 1 year
  Residual volume (RV) (% of predicted) from pre-intervention to follow up
exercise tolerance | 1 year
  Change in the 6 minute walking test from pre-intervention to follow up
Sleepiness evaluation | 1 year
  Epworth sleepiness scale is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'.
  Comparation of patient score from pre-intervention to follow up
acute respiratory exacerbations | 1 year
  Frequency of acute exacerbations of COPD requiring addition of antibiotics and or steroids and or hospital admission
Compliance to PAP | 1 year
  median hours of compliance per night
PAP usage | 1 year
  percentage of days of use per month
Dyspnoea evaluation | 1 year
  The mMRC Dyspnea Scale quantifies disability attributable to breathlessness and is useful for baseline dyspnea characterization in patients with respiratory diseases. The score can range from 0 to 4. The higher the mMRC score the higher the dyspnea.
  Comparation of patient score from pre-intervention to follow up
Symptoms of COPD | 1 year
  COPD Assessment test
Apneia/Hiponeia Index | 1 year
  Number of Residual AHI/per hour
nocturnal hypoventilation | 1 year
  ∆PtcCO2<10mmHg during night from pre-intervention to follow up

IPD SHARING:
Plan to Share IPD: Undecided